CLINICAL TRIAL: NCT05520450
Title: Telematic Support Group in the Care of Domiciliary Patients With Feelings of Loneliness and Social Isolation: a Social Study
Brief Title: Telematic Support Group in Patients With Feelings of Loneliness and Social Isolation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Laura Comendador-Vazquez, Principal Investigator, Corporacion Parc Tauli
Other Study IDs: 2022/3009
Record Dates: First submitted 2022-07-12; First posted 2022-08-30 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Social Isolation; Loneliness
Keywords: Social Isolation; Loneliness; Domiciliary patients; Support group; Telematic
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention group: Recruitment will be based on consecutive patients receiving regular home care in the ATDOM Programme by the Primary Care Team, with prior informed consent.
  Interventions: Behavioral: Telematic support group

INTERVENTIONS:
Behavioral: Telematic support group — The participation of each patient in the study has been established for 4 months; the first and last months correspond to the evaluation phase, the remaining two months are for the intervention. A total of 7 group sessions of 90 minutes duration and weekly frequency are scheduled, carried out via telematics and conducted by an emotional well-being professional, a nurse and a social worker. In this context, it is guaranteed that patients will receive the care, visits and treatments usually used for people who have presented their clinical situation. The only difference between participating in the intervention and not participating in the intervention is the participation in a telematic support group and some additional assessments, i.e. not routinely carried out, which are part of this project. The intervention will be carried out in a group format, with a maximum of 12 patients per session.

SUMMARY:
Loneliness can have negative consequences, both physically and psychologically. The aim of this study is to evaluate the effects of a telematic group intervention in reducing feelings of loneliness and social isolation, as well as improving the emotional well-being of people in home care. The sample is made up of patients aged 60 to 99 years resident in Sabadell health area who receive regular home care in the ATDOM Programme by the Primary Care Team of the Corporació Sanitària Parc Taulí, who agree to participate in the study and meet the eligibility criteria. The study includes clinical assessments, emotional well-being, social support and satisfaction with the intervention.

DETAILED DESCRIPTION:
Loss of autonomy, cognitive impairment and fragility of health can lead to a complex social situation and isolation. Loneliness has been defined as the aversive state that accompanies the perception of a deficit in the quality or quantity of social relationships. It is relevant to conceive loneliness as a complex, diverse and plural phenomenon that requires tools for its detection, understanding and accompaniment during the intervention process. The importance of acting on unwanted loneliness is reflected in the consequences for physical and psychological health. In the long term, chronic and unwanted subjective loneliness leads to consequences such as poorer objective and subjective physical health, increased morbidity and mortality, a risk factor for the development of cognitive impairment, as well as an association with lower self-esteem and sense of identity. The present research study aims to investigate the feasibility of a telematic group intervention in reducing feelings of loneliness and social isolation, as well as improving the emotional well-being of people in home care. A pilot clinical trial with a pre-post intrasubject design will be carried out. The sample is made up of patients aged 60 to 99 years resident in the Sabadell 4B health area who receive regular home care in the ATDOM Programme by the Primary Care Team of the Corporació Sanitària Parc Taulí, who agree to participate in the study and meet the eligibility criteria. The intervention is developed through participation in a telematic support group of 7 sessions of 90 minutes distributed over 2 months, establishing a pre-post intervention evaluation. The study includes clinical assessments, emotional well-being, social support and satisfaction with the intervention. Quantitative variables will be analysed using the non-parametric Wilcoxon signed-rank test. For a more precise interpretation of the relevance of the results in each domain assessed, effect sizes will be calculated for pre-post changes, using Cohen's d. A qualitative analysis of satisfaction with the intervention will also be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 60-99 years.
* Voluntary signature of informed consent.
* Presence of feelings of loneliness and social isolation, self-reported or detected through information from third parties.
* Mobile device with internet connection and basic skills to operate it.
* Literacy: knowing how to read and write.
* People with low psychopathological complexity. The definition is established in patients with mental disorders of low complexity, at a syndromic level related to anxiety and depression. In the absence of difficulties in management, torpid evolution or clarifying clinical need.
* Motivation, attitude and ability to work in a group.
* Receptive attitude to learning new skills and sharing experiences.

Exclusion Criteria:

* People in temporary home care for less than one month (traumatisms, surgery, hospital discharges with a moderate degree of dependency, rehabilitation treatments or therapies).
* Presence of legal incapacitation, not related to a physical level. People with an inability to make decisions due to their mental or intellectual incapacity.
* Comorbidity with disorders incompatible with treatment: moderate or severe cognitive impairment, alterations in verbal communication, severe vision loss or hearing loss.

Ages: 60 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with chronic, degenerative and/or incapacitating pathologies or with unfavourable biopsychosocial characteristics; social isolation, advanced age, autonomy deficits or architectural barriers. Patients aged 60 to 99 years resident in the Sabadell 4B health area who receive regular home care in the ATDOM Programme by the Primary Care Team of the Corporació Sanitària Parc Taulí, who agree to participate in the study and meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change in baseline for loneliness compared to post-intervention | In total, 2 assessments will be carried out. The assessments will take place before and after the intervention, at 4 months. The assessments will last 30 minutes.
  UCLA Loneliness Scale version 3. It will be used to quantify the level of subjective loneliness. It consists of 20 items, which are answered on a 4-point Likert scale (1 = "never" and 4 = "always"). There are no cut-off points; higher scores indicate greater severity of loneliness.
Change in baseline for social isolation compared to post-intervention | In total, 2 assessments will be carried out. The assessments will take place before and after the intervention, at 4 months. The assessments will last 30 minutes.
  OSLO 3 Scale. It will be used to measure perceived social support. It consists of 3 items. Scores between 3 and 8 show poor social support; between 9 and 11 medium social support; between 12 and 15 high social support.
Change in baseline for anxiety and depression compared to post-intervention | In total, 2 assessments will be carried out. The assessments will take place before and after the intervention, at 4 months. The assessments will last 30 minutes.
  Goldberg Anxiety and Depression Scale (EADG). It will be used to quantify the severity of anxiety and depression symptoms. It consists of 18 items measured with dichotomous responses. It contains two subscales, with 9 questions each: anxiety subscale and depression subscale. The first 4 questions of each subscale (questions 1-4) and (questions 10-13) respectively, act as a precondition to determine whether the rest of the questions should be answered. The cut-off points are 4 or more for the anxiety subscale and 2 or more for the depression subscale. Higher scores indicate greater severity of symptoms.

SECONDARY OUTCOMES:
Change in baseline for feasibility of the intervention compared to post-intervention | The assessments will take place after the intervention, at 4 months. The assessments will last 30 minutes.
  Debriefing session with the research team at the end of the intervention. These will be used for qualitative assessment of the feasibility of the intervention: measured by the total number of attendances and absences of the participants in each session.
Change in baseline for satisfaction of the intervention compared to post-intervention | The assessments will take place after the intervention, at 4 months. The assessments will last 30 minutes.
  Debriefing session with the research team at the end of the intervention. These will be used for qualitative assessment of the satisfaction of the intervention: satisfaction with the intervention by the professionals and patients.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Comendador Vazquez, master, Principal Investigator — Corporacion Parc Tauli
Locations (1):
- Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
There is no a plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Sander R. Preventing social isolation and loneliness among older people: a systematic review of health promotion interventions. Nurs Older People. 2005 Mar 1;17(1):40. doi: 10.7748/nop.17.1.40.s11. PMID 27736564
- [Background] Cohen-Mansfield J, Hazan H, Lerman Y, Shalom V. Correlates and predictors of loneliness in older-adults: a review of quantitative results informed by qualitative insights. Int Psychogeriatr. 2016 Apr;28(4):557-76. doi: 10.1017/S1041610215001532. Epub 2015 Oct 1. PMID 26424033
- [Background] Bermeja AI, Ausin B. [Programs to combat loneliness in the institutionalised elderly: A review of the scientific literature]. Rev Esp Geriatr Gerontol. 2018 May-Jun;53(3):155-164. doi: 10.1016/j.regg.2017.05.006. Epub 2017 Nov 1. Spanish. PMID 29100718
- [Background] Courtin E, Knapp M. Social isolation, loneliness and health in old age: a scoping review. Health Soc Care Community. 2017 May;25(3):799-812. doi: 10.1111/hsc.12311. Epub 2015 Dec 28. PMID 26712585
- [Background] Domenech-Abella J, Lara E, Rubio-Valera M, Olaya B, Moneta MV, Rico-Uribe LA, Ayuso-Mateos JL, Mundo J, Haro JM. Loneliness and depression in the elderly: the role of social network. Soc Psychiatry Psychiatr Epidemiol. 2017 Apr;52(4):381-390. doi: 10.1007/s00127-017-1339-3. Epub 2017 Feb 2. PMID 28154893
- [Background] Masi CM, Chen HY, Hawkley LC, Cacioppo JT. A meta-analysis of interventions to reduce loneliness. Pers Soc Psychol Rev. 2011 Aug;15(3):219-66. doi: 10.1177/1088868310377394. Epub 2010 Aug 17. PMID 20716644
- [Background] Morris SB, DeShon RP. Combining effect size estimates in meta-analysis with repeated measures and independent-groups designs. Psychol Methods. 2002 Mar;7(1):105-25. doi: 10.1037/1082-989x.7.1.105. PMID 11928886
- [Background] Syed Elias SM, Neville C, Scott T. The effectiveness of group reminiscence therapy for loneliness, anxiety and depression in older adults in long-term care: a systematic review. Geriatr Nurs. 2015 Sep-Oct;36(5):372-80. doi: 10.1016/j.gerinurse.2015.05.004. Epub 2015 Jun 19. PMID 26099638